CLINICAL TRIAL: NCT05315752
Title: Changes in Body Fat and Morphologic Characteristics Associated With Obstructive Sleep Apnea (OSA) Resolution After Bariatric Surgery
Brief Title: Changes in Body Fat and Morphologic Characteristics Associated With OSA Resolution After Bariatric Surgery
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire Saint Pierre (Other)
Responsible Party: Principal Investigator, Marie Bruyneel, Head of pneumology department, Centre Hospitalier Universitaire Saint Pierre
Other Study IDs: IO-BRUY-CE/220209
Record Dates: First submitted 2022-03-30; First posted 2022-04-07 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Obesity; Obstructive Sleep Apnea
MeSH Terms: conditions — Obesity; Sleep Apnea, Obstructive | interventions — Bariatric Surgery

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Bariatric surgery — Bariatric surgery includes (but is not limited to)
  * Gastric bypass: surgical bypass of the entire stomach, duodenum and approximately 1 m of the proximal small intestine
  * Sleeve: a large part of the stomach is removed laparoscopically, the open vertical edges are put back in place to leave a sleeve-like tube.
  Bariatric surgery is considered a treatment option
  * for patients with a BMI >40 kg/m 2 , assuming the patient has previously participated successfully in a group weight management programme (weight loss >7%) or
  * for patients with a BMI of 35-40 kg/m 2 when the obesity is associated with type 2 diabetes or hypertension, or OAS (with CPAP therapy) or severe musculoskeletal disease

SUMMARY:
Prospective study with inclusion of bariatric surgery candidates with diagnosed Obstructive Sleep Apnea and requiring treatment with Continuous Positive Air Pressure, aiming to evaluate at 2-6-12 months after bariatric surgery whether the relationship between biometric changes (reduction in neck circumference, height, waist/hip ratio, and fat and lean mass) and the resolution of OSA is better than the relationship between these biometric changes and BMI reduction.

DETAILED DESCRIPTION:
Investigators are concerned about the high prevalence of Obstructive Sleep Apnoea syndrome (OSA) in the bariatric population. Postoperatively, there is a high rate of recovery from OSA. Indeed, investigators know from previous reports that weight loss is a very effective, but time consuming, strategy for treating OSA. Patients are therefore treated with CPAP (Continuous Positive Airway Pressure) while waiting for weight loss. In a recent meta-analysis, which focused on the effect of weight loss achieved through lifestyle interventions in 618 overweight and obese patients, the apnea-hypopnea index (AHI) decreased by an amount of 16/h for an average weight loss of 14 kg (1). However, the majority of patients are not able to maintain weight loss in the long term, and weight gain is associated with recurrence/aggravation of OSAS (2). Nowadays, bariatric surgery is a common strategy to achieve sustained and significant weight loss in obese patients. Sarkhosh et al. examined the impact of bariatric surgery (restrictive procedures, with a mild malabsorption component, or largely malabsorptive procedures) on sleep apnoea in 13,900 patients. Depending on the procedure, improvement or resolution of OSAS was achieved in 78-90% of patients (3).

Prospective longitudinal postoperative follow-up study : inclusion of patients who had scheduled bariatric surgery, diagnosed with OSA, AHI > 15 (polysomnography), treated with self-controlled CPAP (APAP), under remote monitoring;

Baseline measures:

1. Anthropometric characteristics: body mass index (BMI), neck circumference, waist/hip ratio, fat mass + lean mass (bioelectrical impedance measurements),
2. APAP treatment characteristics, mean APAP pressure, 95th percentile APAP pressure, APAP adherence.

Follow-up:

1. The 2-month follow-up: body mass index (BMI), neck circumference, waist/hip ratio, fat mass + fat-free mass (bioelectrical impedance measurements), mean APAP pressure, 95th percentile APAP pressure, APAP adherence. To assess potential regression of OSA with weight loss: home polygraphy after 4 nights off APAP (4).
2. Six-month and 12-month follow-up: same as at 2 months. Follow-up stops in case of a polygraph showing an AHI <10, allowing APAP treatment to be stopped.

ELIGIBILITY:
Inclusion Criteria:

Any informed person who is

* eligible for bariatric surgery: with severe obesity (BMI≥35-40) or morbid obesity (BMI≥40), with co-morbidities, who have not lost enough weight with prior lifestyle adaptations (balanced diet, physical activity) AND
* with diagnosed obstructive sleep apnoea (OSA) (AHI > 15/hr on polysomnography) AND
* requiring treatment with Continuous Positive Air Pressure (CPAP)

Exclusion Criteria:

* Cognitive impairment - language barrier

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible patients from CHU St Pierre hospital setting
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-04-22 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Comparison of (1) the relationship between waist circumference changes and resolution of obstructive sleep apnea and (2) the relationship between the changes in waist circumference and BMI | 2 months
  Comparison of (1) the correlation between waist circumference reduction and resolution of OAS (AHI<10/hour on polysomnography) and (2) the correlation between waist circumference reduction and BMI reduction
Comparison of (1) the relationship between waist circumference changes and resolution of obstructive sleep apnea and (2) the relationship between the changes in waist circumference and BMI | 6 months
  Comparison of (1) the correlation between waist circumference reduction and resolution of OAS (AHI<10/hour on polysomnography) and (2) the correlation between waist circumference reduction and BMI reduction
Comparison of (1) the relationship between waist circumference changes and resolution of obstructive sleep apnea and (2) the relationship between the changes in waist circumference and BMI | 12 months
  Comparison of (1) the correlation between waist circumference reduction and resolution of OAS (AHI<10/hour on polysomnography) and (2) the correlation between waist circumference reduction and BMI reduction

SECONDARY OUTCOMES:
Comparison of (1) the correlation between neck circumference reduction and OAS resolution and (2) the correlation between neck circumference reduction and BMI reduction | 2 months
  Comparison of (1) the correlation between neck circumference reduction and OAS resolution (AHI<10/hour on polysomnography) and (2) the correlation between neck circumference reduction and BMI reduction
Comparison of (1) the correlation between neck circumference reduction and OAS resolution and (2) the correlation between neck circumference reduction and BMI reduction | 6 months
  Comparison of (1) the correlation between neck circumference reduction and OAS resolution (AHI<10/hour on polysomnography) and (2) the correlation between neck circumference reduction and BMI reduction
Comparison of (1) the correlation between neck circumference reduction and OAS resolution and (2) the correlation between neck circumference reduction and BMI reduction | 12 months
  Comparison of (1) the correlation between neck circumference reduction and OAS resolution (AHI<10/hour on polysomnography) and (2) the correlation between neck circumference reduction and BMI reduction
Comparison of (1) the correlation between hip circumference reduction and OAS resolution and (2) the correlation between hip circumference reduction and BMI reduction | 2 months
  Comparison of (1) the correlation between hip circumference reduction and OAS resolution (AHI<10/hour on polysomnography) and (2) the correlation between hip circumference reduction and BMI reduction
Comparison of (1) the correlation between hip circumference reduction and OAS resolution and (2) the correlation between hip circumference reduction and BMI reduction | 6 months
  Comparison of (1) the correlation between hip circumference reduction and OAS resolution (AHI<10/hour on polysomnography) and (2) the correlation between hip circumference reduction and BMI reduction
Comparison of (1) the correlation between hip circumference reduction and OAS resolution and (2) the correlation between hip circumference reduction and BMI reduction | 12 months
  Comparison of (1) the correlation between hip circumference reduction and OAS resolution (AHI<10/hour on polysomnography) and (2) the correlation between hip circumference reduction and BMI reduction
Comparison of (1) the correlation between lean mass reduction and OAS resolution and (2) the correlation between lean mass reduction and BMI reduction | 2 months
  Comparison of (1) the correlation between lean mass reduction and OAS resolution (AHI<10/hour on polysomnography) and (2) the correlation between lean mass reduction and BMI reduction
Comparison of (1) the correlation between lean mass reduction and OAS resolution and (2) the correlation between lean mass reduction and BMI reduction | 6 months
  Comparison of (1) the correlation between lean mass reduction and OAS resolution (AHI<10/hour on polysomnography) and (2) the correlation between lean mass reduction and BMI reduction
Comparison of (1) the correlation between lean mass reduction and OAS resolution and (2) the correlation between lean mass reduction and BMI reduction | 9 months
  Comparison of (1) the correlation between lean mass reduction and OAS resolution (AHI<10/hour on polysomnography) and (2) the correlation between lean mass reduction and BMI reduction

CONTACTS AND LOCATIONS:
Locations (2):
- Belgium (2):
  - CHU St Pierre, Brussels
  - Ionela Bold, Brussels